CLINICAL TRIAL: NCT03786861
Title: Corneal Wavefront Guided Versus Aberration Free Transepithelial Photorefractive Keratectomy in Myopic Patients With High Pre-existing Corneal Higher Order Aberrations
Brief Title: Corneal WFG Versus AF Trans PRK in Myopic Patients With High Corneal HOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Amin Faisal Ellakwa, assistant professor, Menoufia University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Al Hekma Center
Record Dates: First submitted 2018-09-02; First posted 2018-12-26 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Myopia
Keywords: aberration free; corneal wavefront guided; higher order aberrations; photorefractive keratectomy.
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 42 eyes in aberration free group (Active Comparator): TransPRK was performed to eligible myopic patients with or without astigmatism with corneal HOAs ≥ 0.35 µ utilizing aberration free in aberration free group provided by ORKCAM software (SCHWIND eye-tech-solutions, Kleinostheim, Germany)
  Interventions: Procedure: corneal WFG group; Procedure: aberration free group
- 24 eyes in corneal WFG group (Active Comparator): TransPRK was performed to eligible myopic patients with or without astigmatism with corneal HOAs ≥ 0.35 µ utilizing corneal WFG patterns in corneal WFG group provided by ORKCAM software (SCHWIND eye-tech-solutions, Kleinostheim, Germany)
  Interventions: Procedure: corneal WFG group; Procedure: aberration free group

INTERVENTIONS:
Procedure: corneal WFG group — TransPRK using ESIRIS flying spot excimer laser system (SCHWIND AMARIS®500E, SCHWIND eye-tech-solutions, Kleinhostheim, Germany), with 500 Hz repetition rate for faster treatments and scanning spots and with smart pulse technology. Eye-tracking during laser ablation was achieved using a 1050 Hz infrared eye tracker centered on the pupil. Static cyclotorsion control (SCC) compensation was obtained for all patients in corneal WFG group.
Procedure: aberration free group — TransPRK was performed to eligible myopic patients with or without astigmatism with corneal HOAs ≥ 0.35 µ utilizing aberration free patterns provided by ORKCAM software (SCHWIND eye-tech-solutions, Kleinostheim, Germany)

SUMMARY:
compare the efficacy, safety and predictability of corneal wavefront guided (WFG) and aberration free ablation in single-step transepithelial photorefractive keratectomy (TransPRK) in myopic patients with high pre-existing corneal higher order aberrations (HOAs).

DETAILED DESCRIPTION:
Objectives:to compare the efficacy, safety and predictability of corneal wavefront guided (WFG) and aberration free ablation in single-step transepithelial photorefractive keratectomy (TransPRK) in myopic patients with high pre-existing corneal higher order aberrations (HOAs).

Background: Corneal WFG and aberration free treatments have been proposed as methods to achieve better visual, refractive, and optical outcomes.

Methods: prospective case series was conducted in El-Hekma Eye-LASIK center, Menoufia governorate, Egypt during the period from January 2017 to December 2017. TransPRK was performed to eligible myopic patients with or without astigmatism with corneal HOAs ≥ 0.35 µ utilizing either aberration free or corneal WFG patterns provided by ORKCAM software (SCHWIND eye-tech-solutions, Kleinostheim, Germany). Uncorrected distance visual acuity (UDVA), manifest and cycloplegic refractions, best spectacle corrected distance visual acuity (CDVA), thorough slit lamp examination and corneal topography were assessed and repeated six months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Myopic patients with or without astigmatism

Exclusion Criteria:

* severe dry eye,
* blepharitis,
* corneal disease,
* contact lens warpage,
* cataract,
* uveitis
* posterior segment anomalies involving the macula or optic nerve
* systemic conditions; diabetes mellitus, connective tissue disease, pregnancy or nursing. Also, any patient who had previous ocular surgery including keratorefractive surgery was excluded

Ages: 21 Years to 52 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — patients 21 years or older with stable refraction for more than 1 year
Enrollment: 33 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
corneal wavefront customized treatments and aberration free aspheric treatments | 1year
  procedure was labeled successful if achieved the desired outcomes in terms of efficacy and safety. Efficacy index was defined as the ratio between the postoperative UDVA to the preoperative CDVA while safety index was defined as the ratio between the postoperative CDVA and the preoperative CDVA. Efficacy index around 1 and safety index more than 1 were desired. Failure was considered when the above outcomes failed to be achieved along with persistence or development of any of the following complications at 6 month postoperative follow up; corneal haze, persistent epithelial defects, ectasia, sterile infiltrate, infectious keratitis, central toxic keratopathy and steroid induced complications

IPD SHARING:
Plan to Share IPD: No